# USEFULNESS OF MULTIMODAL INTRAOPERTIVE NEUROPHYSIOLOGIC MONITORING DURING DIFFERENT NEUROSURGICAL OPERATIONS

**NCT** number: not available

**Document Date: 18 November 2021** 

## Statistical analysis of the data

Data were fed to the computer and analyzed using the IBM SPSS software package version 20.0. (Armonk, NY: IBM Corp) Qualitative data were described using number and percent. The Shapiro-Wilk test was used to verify the normality of the distribution, and quantitative data were described using range (minimum and maximum), mean, standard deviation, median, and interquartile range (IQR). The significance of the results was determined at the 5% level.

#### 1 - Chi-square test

For categorical variables, we compared different groups.

#### 2 - Fisher's Exact or Monte Carlo correction

Correction for chi-square when more than 20% of the cells have expected count less than 5

#### 3 - Sensitivity

 $\frac{TP}{TP + FN} \times 100$ Positivity in diseased patients, expressed as percent =

#### 4 - Specificity

Negativity in non-diseased subjects, expressed as percent =  $\frac{TN}{FP+TN} \times 100$ 5 - Positive Predictive value (PDF)

### 5 - Positive Predictive value (PPV)

Percent of subjects with positive results who are diseased =  $\frac{1P}{TP + FP} \times 100$ 

#### 6 – Negative Predictive value (NPV)

Percent of subjects with negative test results who are non-diseased

$$= \frac{TN}{TN + FN} \times 100$$